CLINICAL TRIAL: NCT03279367
Title: Objective Response Detection to Natural Speech Stimuli for Optimisation of Hearing Aid Fitting Evaluation
Brief Title: Optimisation of Hearing Aid Fitting
Status: Completed | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Royal Berkshire NHS Foundation Trust (Other Government); University of Manchester (Other); Imperial College London (Other); Engineering and Physical Sciences Research Council, UK (Other)
Responsible Party: Sponsor
Other Study IDs: 30123
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss; Hearing Abnormality
Keywords: Hearing Loss; Hearing Abnormality
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hearing Impaired: Participants will be asked to wear an electro-encephalography (EEG) cap for measurement of brain activity whilst listening to speech stimuli. The speech stimuli will be presented through a loudspeaker positioned 1 meter in front of the participant. Participants will be asked to listen to the speech stimuli when using and without using their hearing aid. They will be asked to pay attention to the speech stimuli. This will be assured by asking them to answer questions related to the speech stimulus at random intervals. Subjects will also go through standard clinical procedures for assessing their hearing function and hearing aid setup.
  Interventions: Diagnostic Test: Objective speech response detection

INTERVENTIONS:
Diagnostic Test: Objective speech response detection — Changes in brain activity when a speech stimulus is presented will be measured using electro-encephalography (EEG)

SUMMARY:
This study aims to explore if objective brain responses to speech stimuli (words and running speech) can be used to evaluate hearing aid fitting in adults. Objective brain responses would be beneficial, as they could be used to evaluate hearing with people who are incapable or unwilling to provide subjective responses. The study aims to determine if EEG responses to speech sounds are sensitive to the effects of hearing aids for hearing aid users. Secondary, the study will look into the need for using speech stimuli in order to obtain more robust responses compared to current clinical standards.

DETAILED DESCRIPTION:
The research questions addressed are as follows

1. Are speech-evoked objective brain responses sensitive to hearing aid amplification?
2. Are speech-evoked brain responses sensitive to distortions in speech and can hearing aid amplification resolve issues with brain responses to distorted speech?
3. Which tests are optimal for detection of objective brain responses to speech?
4. Are realistic speech stimuli (words or running speech) able to robustly detect brain responses compared to current clinical standards (clicks and tones)? The study will be carried out on a group of mildly to moderately hearing impaired subjects between the age of 18 and 70. Subjects will be recruited from the Royal Berkshire NHS Foundation Trust, where the research will be conducted. Participants will have their hearing function and hearing aid fitting checked as described in the design and methodology section of this proposal. During the experiment, participants will be asked to listen to speech sounds presented from a loudspeaker at comfortable listening levels. The responses will be measured with the participant wearing and not wearing hearing aids. Additionally, participants will perform a behavioural task for perception of speech. Participants will be asked to attend 2 sessions of 2 hours. Data collection will run over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 18 and 70 years old
* Native English speakers
* Have mild to moderate hearing loss in their better ear measured using current clinical standards
* Routine hearing aid users

Exclusion Criteria:

* Clinical observation indicates the presence of ear infections or an occluded ear canal on the day of testing
* Subjects with recent ear surgery (within a month before the day of testing)
* Subjects who are taking substances that could affect brain responses (e.g. medication for the treatment of depression)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be included if they are between 18 and 70 years old, are native English speakers and have mild to moderate hearing loss in their better ear measured using current clinical standards. They will be identified from their medical records of the Royal Berkshire NHS Foundation Trust by the Co-Investigators who are trained and qualified clinical audiologists at the Trust. Subjects will be routine hearing aid users.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Objective response detection | Immediate
  Detection success rate and time for obtaining a brain response to the sound stimuli.

SECONDARY OUTCOMES:
Improved statistical test | Immediate
  Hotelling's T2 test to objectively determine the presence of a response compared to background noise.
Stimulus reconstruction | Immediate
  Correlation test to determine the accuracy of the estimated speech stimulus using the decoder compared to the presented speech stimulus for running speech.
  Detection of auditory brainstem and auditory steady state potential characteristic peaks and troughs for responses to click and tone stimuli, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Bell, Dr, Principal Investigator — University of Southampton
Locations (1):
- Royal Berkshire NHS Foundation Trust, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be collected and stored in Pure/ePrints at the University of Southampton along with a metadata file describing the procedure and providing participant demographics such as age and gender. Anonymised data will also be stored on password-protected University computers and backed up on password-protected hard drives. Anonymised data will be kept available for public access (for research and teaching purposes) under guidelines of the University of Southampton for at least 10 years. Clear information regarding the storage and possible reuse of anonymized data will be given to the participant prior to the experiment. Participants will have the possibility to opt out of this data sharing policy.

REFERENCES:
- [Result] Vanheusden FJ, Kegler M, Ireland K, Georga C, Simpson DM, Reichenbach T, Bell SL. Hearing Aids Do Not Alter Cortical Entrainment to Speech at Audible Levels in Mild-to-Moderately Hearing-Impaired Subjects. Front Hum Neurosci. 2020 Apr 3;14:109. doi: 10.3389/fnhum.2020.00109. eCollection 2020. PMID 32317951
- [Result] Vanheusden FJ, Chesnaye MA, Simpson DM, Bell SL. Envelope frequency following responses are stronger for high-pass than low-pass filtered vowels. Int J Audiol. 2019 Jun;58(6):355-362. doi: 10.1080/14992027.2018.1562243. Epub 2019 Jan 24. PMID 30675827
- [Result] Vanheusden FJ, Bell SL, Chesnaye MA, Simpson DM. Improved Detection of Vowel Envelope Frequency Following Responses Using Hotelling's T2 Analysis. Ear Hear. 2019 Jan/Feb;40(1):116-127. doi: 10.1097/AUD.0000000000000598. PMID 29757799

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03279367/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03279367/ICF_001.pdf